CLINICAL TRIAL: NCT02873143
Title: 5 Year Follow-up of Adolescents With Knee Pain - a Prospective Cohort Study of 504 Adolescents
Brief Title: 5 Year Follow-up of Adolescents With Knee Pain
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Research Unit for General Practice in Aalborg (Other); University of Southern Denmark (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Senior researcher, Aalborg University
Other Study IDs: 2011-0020
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Patellofemoral Pain Syndrome; Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The APA2011 cohort: In September 2011, students at 4 upper secondary schools in Aalborg were invited to answer an online questionnaire and to be part of the APA2011 cohort. From 2846 potential responders, 2200 adolescents responded to the questionnaire, corresponding to a response rate of 77%. A total of 504 adolescents indicating knee pain at least monthly were successfully contacted (a response rate of 83% of those who reported their telephone numbers) and were asked standardized questions on the telephone. This forms the cohort of 504 adolescents with knee pain. In addition a random selected group of adolescents without knee pain in 2011 will be contacted and asked the same questions as those with knee pain.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The prevalence of adolescent knee pain is 33%, and patellofemoral pain (PFP) is the most common diagnosis with a nontraumatic onset. The 5-year prognosis of adolescent PFP compared with other types of knee pain is unknown.

In 2011, a cohort of 2200 adolescents aged 15 to 19 years answered an online questionnaire on musculoskeletal pain. Of these, 504 reported knee pain, and 153 of these were clinically diagnosed with PFP. Now, after 5 years, the 504 adolescents, as well as 252 randomly selected adolescents who did not report knee pain in 2011, will be contacted again to gain insights into their prognosis.

ELIGIBILITY:
From the 504, 153 were diagnosed with PFP, the criteria for which included:

- insidious onset of anterior knee or retropatellar pain for longer than 6 weeks that was provoked by at least 2 of the following: prolonged sitting or kneeling, squatting, running, hopping, or stair climbing; tenderness on palpation of the patella; pain when stepping down; or double-leg squatting.

Exclusion criteria were:

* concomitant injury or pain from the hip, lumbar spine, or other knee structures
* self-reported patellofemoral instability
* knee joint effusion.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In September 2011, students at 4 upper secondary schools in Aalborg were invited to answer an online questionnaire and to be part of the APA2011 cohort. From 2846 potential responders, 2200 adolescents responded to the questionnaire, corresponding to a response rate of 77%. A total of 504 adolescents indicating knee pain at least monthly were successfully contacted (a response rate of 83% of those who reported their telephone numbers) and were asked standardized questions on the telephone. This forms the cohort of 504 adolescents with knee pain. In addition a random selected group of adolescents without knee pain in 2011 will be contacted and asked the same questions as those with knee pain.
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Knee pain during the last week | 5 years
  All subjects are asked if they experienced knee pain during the last week

SECONDARY OUTCOMES:
Knee pain during the last 30 days | 5 years
  Did you experience knee pain during the last 30 days?
Frequency of knee pain | 5 years
  Frequency of knee pain divided into (almost daily, several times per week, weekly, monthly, rarely, never
When did your knee pain resolve | 5 years
Pain in other regions of the body | 5 years
Seeking medical attention for your knee pain | 5 years
Previous treatments for your knee pain | 5 year
Use of pain medication | 5 years
Worst pain last week | 5 years
  Measured on a numeric rating scale
Knee Injury and Osteoarthritis Outcome score | 5 years
Health-related quality of life | 5 years
  Measure with the EQ-5D-3L
The influence of knee pain on choice of activity level, mood, choice of education and professional career | 5 years
Physical activity level | 5 years
  Measured with the IPAQ
Number of sports participation per week | 5 years
The effect of knee pain on sports participation | 5 years
Self-reported sleep problems | 5 years
  Assessed by asking three questions related to: trouble falling asleep, wake several times per night and trouble staying asleep.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rathleff MS, Holden S, Straszek CL, Olesen JL, Jensen MB, Roos EM. Five-year prognosis and impact of adolescent knee pain: a prospective population-based cohort study of 504 adolescents in Denmark. BMJ Open. 2019 May 28;9(5):e024113. doi: 10.1136/bmjopen-2018-024113. PMID 31142518